CLINICAL TRIAL: NCT01233414
Title: Randomized Trial of Parent Training for Young Children With Autism
Acronym: RUBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Emory University (Other); Indiana University (Other); Ohio State University (Other); University of Pittsburgh (Other); University of Rochester (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Denis Sukhodolsky, Assistant Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH081148 (NIH); R01MH081148 (NIH)
Record Dates: First submitted 2010-10-29; First posted 2010-11-03 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Child Development Disorders, Pervasive
Keywords: Pervasive Developmental Disorder; Autism; Children; Behavior Therapy; Aggression; Tantrums; Noncompliance
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autistic Disorder; Aggression; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent Training (Experimental)
  Interventions: Behavioral: Parent Training
- Psychoeducation (Active Comparator)
  Interventions: Other: Psychoeducational Program

INTERVENTIONS:
Behavioral: Parent Training — The Parent Training program will be delivered individually to the parents of study participants. Families will attend up to 13 90-minute treatment sessions over a 24-week period. Topics covered in the program include reinforcement, teaching compliance, and functional communication. The treatment sessions employ direct instruction, review of video-taped examples, practice activities, behavior rehearsal with feedback, and role-playing to accomplish specific skill acquisition. Parents will be given specific homework assignments between sessions.
  Arms: Parent Training
Other: Psychoeducational Program — The Psychoeducational program will be delivered individually to the parents of study participants. Families will attend up to 13 90-minute informational sessions over a 24-week period. The program provides an overview on a variety of topics including the complexities of a PDD diagnosis, co-occurring medical conditions, relevant aspects of child development, use of medications, treatment options for challenging behavior, nutritional issues, and complementary and alternative treatments.
  Arms: Psychoeducation

SUMMARY:
The purpose of this 24 week study is to determine whether a new Parent Training program is effective in reducing disruptive behaviors in young children with pervasive developmental disorders.

DETAILED DESCRIPTION:
Pervasive Developmental Disorders (PDDs) are a group of conditions that includes Autistic Disorder, Asperger's disorder and so called Pervasive Developmental Disorder - Not Otherwise Specified. Children with PDD show delays in speech and language and reduced social interaction. Some children with PDD also have behavior problems, including defiance of rules, aggression, and tantrums. The purpose of this study is to evaluate a new Parent Training program designed to decrease these behavior problems and improve daily living skills.

Following confirmation of eligibility, participants will be randomly assigned to receive either Parent Training or a Psychoeducational Program. The Parent Training program involves specific suggestions about how to deal with behavior problems. The Psychoeducational program covers specific issues related to autism and parenting, including an co-occurring medical conditions and treatment options.

Parents will attend up to 13 one-on-one sessions with a trained therapist over a 24-week period. Participation in the study also involves 2 home visits and 6 monthly assessment visits. The purpose of the assessment visits is to evaluate the child's response to treatment. Evaluations will also be conducted at 3 and 6 months after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autistic Disorder, Pervasive Developmental Disorder, Not Otherwise Specified, or Asperger's Disorder
* Between ages 3 yrs 0 months and 6 yrs 11 months.
* No planned changes in the intensity of current treatment(s)
* Medication free or on stable medication

Exclusion Criteria:

* Diagnosis of Rett's Disorder or Childhood Disintegrative Disorder
* Participation in a structured parent training program in the past 2 years
* Developmental age < 18 months (IQ < 35)

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist Irritability Subscale | Week 24
Home Situations Questionnaire | Week 24

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scales | Week 24
Clinical Global Impressions Improvement Scale | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Scahill, MSN, PhD, Principal Investigator — Emory University; Cynthia Johnson, PhD, Principal Investigator — University of Pittsburgh; Tristram Smith, PhD, Principal Investigator — University of Rochester; Luc Lecavalier, PhD, Principal Investigator — Ohio State University; Naomi Swiezy, PhD, Principal Investigator — Indiana University; Denis Sukhodolsky, PhD, Principal Investigator — Yale University
Locations (6):
- United States (6):
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Rochester, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Aman MG, McDougle CJ, Scahill L, Handen B, Arnold LE, Johnson C, Stigler KA, Bearss K, Butter E, Swiezy NB, Sukhodolsky DD, Ramadan Y, Pozdol SL, Nikolov R, Lecavalier L, Kohn AE, Koenig K, Hollway JA, Korzekwa P, Gavaletz A, Mulick JA, Hall KL, Dziura J, Ritz L, Trollinger S, Yu S, Vitiello B, Wagner A; Research Units on Pediatric Psychopharmacology Autism Network. Medication and parent training in children with pervasive developmental disorders and serious behavior problems: results from a randomized clinical trial. J Am Acad Child Adolesc Psychiatry. 2009 Dec;48(12):1143-54. doi: 10.1097/CHI.0b013e3181bfd669. PMID 19858761
- [Background] Johnson CR, Handen BL, Butter E, Wagner A, Mulick J, Sukhodolsky DG, Williams, S, Swiezy, NA, Arnold LE, Aman MG, Scahill L, Stigler KA, McDougle CJ, Vitiello B, Smith T (2007). Development of a Parent Management Training Program for Children with Pervasive Developmental Disorders. Behav Intervent, 22:1-21.
- [Background] Bearss K, Johnson C, Smith T, Lecavalier L, Swiezy N, Aman M, McAdam DB, Butter E, Stillitano C, Minshawi N, Sukhodolsky DG, Mruzek DW, Turner K, Neal T, Hallett V, Mulick JA, Green B, Handen B, Deng Y, Dziura J, Scahill L. Effect of parent training vs parent education on behavioral problems in children with autism spectrum disorder: a randomized clinical trial. JAMA. 2015 Apr 21;313(15):1524-33. doi: 10.1001/jama.2015.3150. PMID 25898050
- [Derived] Scahill L, Bearss K, Lecavalier L, Smith T, Swiezy N, Aman MG, Sukhodolsky DG, McCracken C, Minshawi N, Turner K, Levato L, Saulnier C, Dziura J, Johnson C. Effect of Parent Training on Adaptive Behavior in Children With Autism Spectrum Disorder and Disruptive Behavior: Results of a Randomized Trial. J Am Acad Child Adolesc Psychiatry. 2016 Jul;55(7):602-609.e3. doi: 10.1016/j.jaac.2016.05.001. Epub 2016 May 7. PMID 27343887